CLINICAL TRIAL: NCT06277505
Title: Efficacy and Safety Evaluation of Prebiotics Combined With Quadruple Probiotics in Improving Functional Constipation: a Prospective Randomized Controlled Open-label Study
Brief Title: Efficacy and Safety Evaluation of Prebiotics Combined With Quadruple Probiotics in Improving Functional Constipation.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023(164)
Record Dates: First submitted 2024-02-18; First posted 2024-02-26 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-03

CONDITIONS: Functional Constipation
Keywords: prebiotics; probiotics; functional constipation; Randomized Controlled Trial
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotics and probiotics，life-style (Experimental): Take 3.5g prebiotic +2g probiotic twice a day before meals; At the same time, lifestyle guidance is given, including adjusting dietary structure, increasing the intake of foods high in dietary fiber and moderate exercise
  Interventions: Combination Product: Take prebiotics and probiotics; Behavioral: lifestyle guidance
- life-style (Other): lifestyle guidance is given, including adjusting dietary structure, increasing the intake of foods high in dietary fiber and moderate exercise
  Interventions: Behavioral: lifestyle guidance

INTERVENTIONS:
Combination Product: Take prebiotics and probiotics — Take 3.5g prebiotic +2g prebiotic twice a day before meals; At the same time, lifestyle guidance is given, including adjusting dietary structure, increasing the intake of foods high in dietary fiber and moderate exercise
  Other Names: behavioral
  Arms: Prebiotics and probiotics，life-style
Behavioral: lifestyle guidance — lifestyle guidance is given, including adjusting dietary structure, increasing the intake of foods high in dietary fiber and moderate exercise

SUMMARY:
In this study, we will evaluate the efficacy of prebiotics combined with quadruple probiotics in the treatment of functional constipation through an open RCT study. The experimental group received lifestyle guidance and combined intervention of prebiotics and quadruple probiotics at the same time. The patients took the combination of prebiotics and probiotics twice a day during the treatment period. The control group received only lifestyle instruction. At the same time, to evaluate the safety of probiotics combined with quadruple probiotics in the treatment of functional constipation, and provide a new treatment plan for clinical treatment of functional constipation.

DETAILED DESCRIPTION:
The purpose of this study is to analyze the intestinal microecology of patients with functional constipation before and after treatment through intestinal microecological intervention, mainly using the combination of probiotics and prebiotics. We will record the patient's stool diary, including bowel movements, stool quality, bowel time, defecation difficulty, emptying sensation, manual operation and medication. At the same time, we will use the Bristol Fecal Traits Scale (BSFS) and the Constipation Patient Self-Rating Scale (PAC-SYM) and Constipation Patient Quality of Life Scale (PAC-QOL) scores completed weekly. In addition, we will monitor indicators of inflammation (IL-1β, IL-6, TNF-alpha) and intestinal barrier function (LPS), neurotransmitter (serotonin, acetylcholine)) to assess constipation improvement in patients with functional constipation.

ELIGIBILITY:
Inclusion Criteria:

1. Age: between 18 and 60 years old
2. Functional constipation was diagnosed using Rome IV criteria.
3. No other relevant medications that may affect the gut microbiota before the start of the experiment
4. Ability to participate
5. Consent to participate in the study

Exclusion Criteria:

1. Organic constipation (such as intestinal obstruction, bowel cancer, etc.)
2. Outlet obstructive constipation
3. Previous abdominal, rectal, or perianal surgery except cholecystectomy, appendectomy, tubal ligation, and cesarean section
4. Patients with constipation-oriented irritable bowel syndrome (IBS-C) or functional abdominal pain syndrome who meet Rome IV criteria
5. a serious mental illness or any medical condition related to it
6. Diseases of the small or large intestine, such as ulcerative colitis and Crohn's disease
7. There are serious important organs such as respiratory, heart, liver, kidney and other functional insufficiency
8. Use probiotics, prebiotics and/or Biostime within 1 month

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in the number of fully autonomous bowel movements per week at the end of treatment | A month after treatment
  Change in the number of fully autonomous bowel movements per week at the end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen Univisity, Xiamen, Fujian, China